CLINICAL TRIAL: NCT07006974
Title: Patients With Left Ventricular Hypertrophy in Syndromic and Metabolic Cardiomyopathy Compared to Hypertrophic Cardiomyopathy: an Age-sex Matched Cohort Study
Brief Title: SMCs With LVH Compared to HCM
Status: Active, not recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-ZDYF-01-4
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Syndromic and Metabolic Cardiomyopathy; Cardiomyopathies
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: SMCs — patients with SMCs

SUMMARY:
The goal of this cohort study is to investigate the clinical characteristics of SMCs and to explore the difference in cardiovascular outcomes in comparison to age-, sex-, and admission year-matched HCM patients. The main question it aims to answer is:

* Do patients with SMCs have higher rates of cardiac outcomes?
* What risk factors do SMCs patients experience a poor prognosis?

ELIGIBILITY:
Inclusion Criteria:

* patients who were diagnosed SMCs or HCM. Gene testing and muscle biopsy were used to confirm the diagnosis of SMCs. The diagnose of HCM was according to the 2024 ESC Guidelines of HCM but without evidence of SMCs.
* complete baseline data
* accessible follow-up data

Exclusion Criteria:

* incomplete baseine data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators identified patients with SMCs by screening the electronic database. Gene testing and muscle biopsy were used to confirm the diagnosis of SMCs. (Part two) Patients with HCMs were included as the controls of SMCs who had LVH and available CMR data in our study. The diagnose of HCM was according to the 2024 ESC Guidelines of HCM but without evidence of SMCs. Controls were matched 1:2 to each case based on sex, age (matched within ± 5 years), and admission year (matched within ± 12 months).
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
primary outcome | 3 years
  a composite of all-cause death, hospitalization for heart failure, myocardial infarction, ischemia or hemorrhagic stroke (excluding transient ischemic attack), other thrombotic events, and modified International Society on Thrombosis and Haemostasis crit

CONTACTS AND LOCATIONS:
Overall Officials: Liang, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided